CLINICAL TRIAL: NCT05855681
Title: Effect Of Strengthening Hip Rotators And Ankle Muscles On Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Osama Mohammed Galal ALSaadawy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004359
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Triple blinded Randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) (assessor by research assistant, patients and statistician)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): patients will receive strengthening exercise for hip rotators and ankle muscles in addition to quadriceps strengthening . stretching exercise for hamstring and calf muscle also will be received
  Interventions: Other: therapeutic exercises
- control group (Other): patients will receive strengthening exercises for quadriceps and stretching exercise for hamstring and calf muscle.
  Interventions: Other: therapeutic exercises

INTERVENTIONS:
Other: therapeutic exercises — strengthening exercise and stretching exercise

SUMMARY:
The goal of this clinical trial is to investigate the effect of adding strengthening exercise for hip rotators and ankle muscles to knee exercises on pain, function, muscles strength , and knee proprioception in patients with knee osteoarthritis.

The main question it aims to answer is:

* What is the effect of adding strengthening exercise for hip rotators and ankle muscles to knee exercises on pain, function, strength of hip rotators and ankle muscles, and knee proprioception in patients with knee osteoarthritis?" Adult male and female diagnosed with unilateral or bilateral knee osteoarthritis, referred from orthopedic surgeons according to inclusion and exclusion criteria will be enrolled in this study, randomly allocated to groups and received exercise for 4 weeks.
* Control group Patients in this group will receive knee exercises in the form of stretching for hamstring and calf. Strengthening exercises in form of strengthening exercise for quadriceps.
* Experimental group In addition to the same knee exercise of control group patients will receive strengthening exercise for hip rotators and ankle muscles.

DETAILED DESCRIPTION:
The purpose of the current study is to investigate the effect of adding strengthening exercise for hip rotators and ankle muscles to knee exercises on pain, function, strength of muscles, and knee proprioception in patients with knee osteoarthritis. Adult male and female diagnosed with unilateral or bilateral knee osteoarthritis, referred from orthopedic surgeons according to inclusion and exclusion criteria will be enrolled in this study, randomly allocated to groups and received exercise for 4 weeks. Control group Patients in this group will receive knee exercises in the form of stretching for hamstring and calf. Strengthening exercises in form of strengthening exercise for quadriceps. Experimental group In addition to the same knee exercise of control group patients will receive strengthening exercise for hip rotators and ankle muscles.

Recruited subjects will be screened with consideration of the inclusion and exclusion criteria. Aim of the study and all testing procedures will be verbally explained for eligible subjects and all relevant questions will be answered. If they agreed to participate in the study, an informed consent will be signed . Then, basic demographic information will be collected and patients will start the test. We will measure pain using visual analogue scale, functional level of the knee using Arabic Knee injury and Osteoarthritis Outcome Score questionnaire, isometric muscle strength of quadriceps, hip external and internal rotators, dorsi flexors, planter flexors, evertors and invertor muscles of ankle will be measured by handheld dynamometer and finally knee proprioception will be measured by assessing joint position sense by digital inclinometer. All these measurements will be done at base line and after (4 week) at the end of the treatment program.

All patients will receive knee exercises according to guidelines and previous studies in the form of strengthening exercises that progress from 50% of the

1. repetition maximum at first 2 week to 70% of 1 repetition maximum at last
2. weeks, and from mild and moderate Thera band resistance in the first 2 weeks to maximum resistance in the last 2 weeks. In addition to knee muscle strengthening exercises,the experimental group will receive hip rotators and ankle muscles strengthening exercises. Passive stretching for hamstring and calf muscles will be done at the end of all exercises. Stretching will be performed three repetitions per session, holding each stretch for 30 seconds, with 10-seconds rest in between. All exercises will be performed for 30 to 45 minutes per session, 3 times per week for 4 weeks (12 sessions).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Knee osteoarthritis with pain for more than 3 months.
2. Age between 40-55 years .
3. BMI 25 - 34.9
4. Kellgren _ Lawrence grad1,2,3 .
5. Subjects must be referred to the outpatient clinic of the faculty of Physical Therapy, Cairo University with a confirmed diagnosis of unilateral or bilateral (knee with primary affection included) knee osteoarthritis and having one or more of the following criteria:

   1. Morning stiffness for less than 30 min.
   2. Crepitus on active knee movement.
   3. Palpable or radiographic bony enlargement.
   4. Tenderness at joint margins or joint line.
6. Knee pain over 30 mm on the Visual analogue scale.

Exclusion Criteria:

- 1- Physical therapy treatment for hip, knee and ankle in the last month. 2-Steroid knee injections in the previous 3 months. 3- hyaluronic acid intraarticular injections in the previous 6 months. 4- History of knee, ankle or hip surgery in the last 2 years. 5- Severe knee malalignment in varus or valgus that requires use of any gait-assistive device.

6- Neurological disease in lower limb 7- Inflammatory arthritis (eg: rheumatoid arthritis). 8- Ankle instability

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
pain level | 4 weeks
  assessed by visual analogue scale
functional level | 4 weeks
  assessed by Knee injury and Osteoarthritis Outcome Score
knee proprioception | 4 weeks
  assessed by joint position sense

SECONDARY OUTCOMES:
Hip internal and external rotator strength | 4 weeks
  assessed by handheld dynamometer
Ankle dorsi flexors, planter flexor, invertor and evertor strength | 4 weeks
  assessed by handheld dynamometer
Quadriceps strength | 4 weeks
  assessed by handheld dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt